CLINICAL TRIAL: NCT00379457
Title: A Protocol For Nonmetastatic Rhabdomyosarcoma [RMS-2005]
Brief Title: Combination Chemotherapy in Treating Young Patients With Nonmetastatic Rhabdomyosarcoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Paediatric Soft Tissue Sarcoma Study Group (Other)
Collaborators: Italian Association for Pediatric Hematology Oncology (Other); Children's Cancer and Leukaemia Group (Other); Dutch Childhood Oncology Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CCLG-EPSSG-RMS-2005; CDR0000508635 (Registry Identifier: PDQ (Physician Data Query)); EU-20639; EUDRACT-2005-000217-35; UKCCSG-RMS-2005
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Sarcoma
Keywords: alveolar childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; childhood malignant mesenchymoma; nonmetastatic childhood soft tissue sarcoma; embryonal childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma; Malignant mesenchymal tumor | interventions — Dactinomycin; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Topotecan; Vincristine; Vinorelbine; Radiotherapy

INTERVENTIONS:
Biological: dactinomycin
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: topotecan hydrochloride
Drug: vincristine sulfate
Drug: vinorelbine tartrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating rhabdomyosarcoma.

PURPOSE: This randomized phase III trial is studying different combination chemotherapy regimens to compare how well they work in treating young patients with nonmetastatic rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Improve the outcome in pediatric patients with low-risk rhabdomyosarcoma (RMS) treated with vincristine and dactinomycin alone.
* Evaluate whether the outcome for older patients with standard-risk RMS with favorable features may be improved/maintained by administering a treatment with limited intensity.
* Evaluate whether chemotherapy intensity for patients with standard-risk RMS can be reduced, by lowering the cumulative dose of ifosfamide.
* Evaluate whether treatment can be reduced in a subgroup of patients with standard-risk RMS arising in an unfavorable site (e.g., parameningeal or other site) but with favorable site and age.
* Compare the value of standard chemotherapy comprising ifosfamide, vincristine, and dactinomycin with vs without doxorubicin (as early intensification in the initial part of treatment) in patients with high-risk RMS.
* Determine the role of low-dose maintenance chemotherapy comprising 6 months of cyclophosphamide and vinorelbine in patients with high-risk RMS.
* Improve the results in patients with poor prognosis (very high-risk) RMS treated with more intensive ifosfamide, vincristine, dactinomycin, and doxorubicin followed by maintenance chemotherapy.

OUTLINE: This is a non-blinded, randomized, prospective, multicenter study. Patients are stratified according to risk group (low risk vs standard risk vs high risk vs very high risk) and participating country.

* Stratum 1 (low-risk group): Patients receive vincristine IV on day 1 in weeks 1-4, 7-10, 13-16, and 19-22 and dactinomycin IV on day 1 in weeks 1, 4, 7, 10, 13, 16, 19, and 22.
* Stratum 2 (standard-risk group): Patients are assigned to 1 of 3 treatment groups according to their standard-risk subgroup.

  * Subgroup B: Patients receive ifosfamide IV over 3 hours on days 1 and 2 in weeks 1, 4, 7, and 10; vincristine IV on day 1 in weeks 1-7, 10, 13, 16, 19, 22, and 25; and dactinomycin IV on day 1 in weeks 1, 4, 7, 10, 13, 16, 19, 22, and 25.
  * Subgroup C: Patients receive ifosfamide IV over 3 hours on days 1 and 2 in weeks 1, 4, and 7; vincristine IV on day 1 in weeks 1-7; and dactinomycin IV on day 1 in weeks 1, 4, and 7. Patients are evaluated for tumor response in week 9. Patients in complete remission (CR) with favorable age and tumor size continue to receive ifosfamide, vincristine, and dactinomycin as above in weeks 10, 13, 16*, 19, 22, and 25. Patients may also undergo radiotherapy beginning in week 13 and continuing for 5-6 weeks. Patients in CR with unfavorable age or tumor size OR in partial remission (PR) (i.e., > 1/3 tumor volume reduction) continue to receive ifosfamide as above in weeks 10 and 16 and vincristine and dactinomycin as above in weeks 10, 13, 16*, 19, 22, and 25. These patients also undergo radiotherapy beginning in week 13 and continuing for 5-6 weeks. Patients with stable or progressive disease in week 9 proceed to second-line therapy and radiotherapy. Patients with residual disease after completion of chemotherapy in week 10 undergo surgical resection followed by ifosfamide, vincristine, and dactinomycin (with or without radiotherapy) as above in weeks 13, 16*, 19, 22, and 25.
  * Subgroup D: Patients receive ifosfamide IV over 3 hours on days 1 and 2 in weeks 1, 4, and 7; vincristine IV on day 1 in weeks 1-7; and dactinomycin IV on day 1 in weeks 1, 4, and 7. Patients are evaluated for tumor response in week 9. Patients in CR or PR continue to receive ifosfamide, vincristine, and dactinomycin as above in weeks 10, 13, 16*, 19, 22, and 25. Patients may also undergo radiotherapy beginning in week 13 and continuing for 5-6 weeks. Patients with stable or progressive disease in week 9 proceed to second-line therapy and radiotherapy. Patients with residual disease after completion of chemotherapy in week 10 undergo surgical resection followed by ifosfamide, vincristine, and dactinomycin (with or without radiotherapy) as above in weeks 13, 16*, 19, 22, and 25.

NOTE: *Dactinomycin may be omitted during radiotherapy in week 16.

* Stratum 3 (high-risk group): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive ifosfamide, vincristine, and dactinomycin as in subgroups C and D of stratum 2. Patients are evaluated for tumor response in week 9. Patients in CR or PR continue to receive ifosfamide, vincristine, and dactinomycin as in subgroups C and D of stratum 2. Patients may also undergo radiotherapy beginning in week 13 and continuing for 5-6 weeks. Patients with stable or progressive disease in week 9 proceed to second-line therapy and radiotherapy. Patients with residual disease after completion of chemotherapy in week 10 undergo surgical resection followed by ifosfamide, vincristine, and dactinomycin (with or without radiotherapy) as above in weeks 13, 16*, 19, 22, and 25.
  * Arm II: Patients receive ifosfamide, vincristine, and dactinomycin as in subgroups C and D of stratum 2. Patients also receive doxorubicin IV over 4 hours on days 1 and 2 in weeks 1, 4, and 7. Patients are evaluated for tumor response in week 9. Patients in CR or PR continue to receive ifosfamide, vincristine, dactinomycin, and doxorubicin as above in week 10 and then ifosfamide, vincristine, and dactinomycin as above in weeks 13, 16*, 19, 22, and 25. Patients may also undergo radiotherapy beginning in week 13 and continuing for 5-6 weeks. Patients with stable or progressive disease in week 9 proceed to second-line therapy and radiotherapy. Patients with residual disease after completion of chemotherapy in week 10 undergo surgical resection followed by ifosfamide, vincristine, and dactinomycin (with or without radiotherapy) as above in weeks 13, 16*, 19, 22, and 25.

NOTE: *Dactinomycin may be omitted during radiotherapy in week 16.

* Maintenance chemotherapy: Patients who remain in CR or with minimal abnormalities on imaging studies after completion of therapy according to their randomized arm (as above) undergo a second randomization. Randomization occurs within 6 weeks after administration of the last course of chemotherapy on arm I or II.

  * Arm I: Patients receive no maintenance chemotherapy.
  * Arm II: Patients receive vinorelbine IV over 5-10 minutes on days 1, 8, and 15 and oral cyclophosphamide once daily on days 1-28. Treatment repeats every 28 days for up to 6 courses.

    * Stratum 4 (very high-risk group): Patients receive ifosfamide, vincristine, and dactinomycin as in subgroups C and D of stratum 2. Patients also receive doxorubicin as in arm II of stratum 3. Patients are evaluated for tumor response in week 9. Patients in CR or PR continue to receive ifosfamide, vincristine, dactinomycin, and doxorubicin as in arm II of stratum 3. Patients may also undergo radiotherapy beginning in week 13 and continuing for 5-6 weeks. Patients with stable or progressive disease in week 9 proceed to second-line therapy and radiotherapy. Patients with residual disease after completion of chemotherapy in week 10 undergo surgical resection followed by ifosfamide, vincristine, and dactinomycin (with or without radiotherapy) as above in weeks 13, 16, 19, 22, and 25. After completion of chemotherapy, patients with a limited quantity of viable tumor proceed to maintenance chemotherapy.
* Maintenance chemotherapy: Patients receive vinorelbine IV over 5-10 minutes on days 1, 8, and 15 and oral cyclophosphamide once daily on days 1-28. Treatment repeats every 28 days for up to 6 courses.

  * Second-line therapy: Patients in any stratum with stable or progressive disease in week 9 receive 1 of 2 second-line therapy regimens.
* Regimen 1: Patients receive topotecan IV on days 1-3 and carboplatin IV on days 4 and 5 in weeks 1 and 4. Patients are then evaluated for tumor response. Patients with good response receive topotecan IV on days 1-3 and cyclophosphamide IV on days 1 and 2 in weeks 7 and 13 and etoposide IV on days 1-3 and carboplatin IV on days 4 and 5 in weeks 10 and 16. Patients with no response receive local therapy or a new chemotherapy regimen.
* Regimen 2: Patients receive doxorubicin IV on day 1 and carboplatin IV on days 1 and 2 in weeks 1 and 4. Patients are then evaluated for tumor response. Patients with good response receive doxorubicin IV on day 1 in weeks 7, 10, 13, and 16; cyclophosphamide IV on days 1 and 2 in weeks 7 and 13; and carboplatin IV on days 1 and 2 of weeks 10 and 16. Patients with no response receive local therapy or a new chemotherapy regimen.

After completion of therapy, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed rhabdomyosarcoma (RMS) or other malignant mesenchymal tumor, including undifferentiated soft tissue sarcoma or ectomesenchymoma

  * Has undergone diagnostic surgery within the past 8 weeks
* Meets criteria for 1 of the following risk groups:

  * Low-risk group

    * Localized nonalveolar RMS at any site
    * Embryonal, spindle cell, or botryoid RMS (favorable pathology)
    * Microscopically completely resected disease (Intergroup Rhabdomyosarcoma Study [IRS] group I)
    * Negative nodes (N0)
    * Tumor size ≤ 5 cm AND age < 10 years (favorable tumor size and age)
  * Standard-risk group, meeting criteria for 1 of the following subgroups:

    * Subgroup B

      * Localized nonalveolar RMS at any site
      * Favorable pathology
      * Microscopically completely resected disease (IRS group I)
      * N0 disease
      * Tumor size > 5 cm OR age ≥ 10 years (unfavorable tumor size or age)
    * Subgroup C

      * Localized nonalveolar RMS in orbit, head and neck nonparameningeal sites, or genitourinary (GU) non bladder prostate (i.e., paratesticular and vagina/uterus) sites (favorable site)
      * Favorable pathology
      * Microscopic residual disease (pT3a) or completely resected disease with nodal involvement (N1) (IRS group II) OR macroscopic residual disease (pT3b) (IRS group III)
      * N0 disease
      * Any tumor size or age
    * Subgroup D

      * Localized nonalveolar RMS in parameningeal sites, extremities, GU bladder prostate sites, or other sites (unfavorable site)
      * Favorable pathology
      * IRS group II or III
      * N0 disease
      * Favorable tumor size and age
  * High-risk group, meeting criteria for 1 of the following subgroups:

    * Subgroup E

      * Localized nonalveolar RMS at unfavorable site
      * Favorable pathology
      * IRS group II or III
      * N0 disease
      * Unfavorable tumor size or age
    * Subgroup F

      * Localized nonalveolar RMS at any site
      * Favorable pathology
      * IRS group I, II, or III
      * Positive nodes (N1)
      * Any tumor size or age
    * Subgroup G

      * Localized alveolar RMS at any site
      * Alveolar RMS, including the solid-alveolar variant (unfavorable pathology)
      * IRS group I, II, or III
      * N0 disease
      * Any tumor size or age
  * Very high-risk group

    * Localized alveolar RMS at any site
    * Unfavorable pathology
    * IRS group I, II, or III
    * N1 disease
    * Any tumor size or age
* Previously untreated disease (except for primary surgery)
* No evidence of metastatic disease

PATIENT CHARACTERISTICS:

* Shortening fraction > 28%
* Ejection fraction > 47%
* No prior cardiac disease
* Renal function must be equivalent to grade 0-1 nephrotoxicity
* No prior malignant tumors
* No pre-existing illness preventing treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-06; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival
Disease-free survival (in patients treated with maintenance chemotherapy)

SECONDARY OUTCOMES:
Overall survival
Progression-free survival
Response rate
Toxicity as measured by NCI-CTC version 3

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Bisogno, MD, Study Chair — Azienda Ospedaliera di Padova; Meriel Jenney, MD, Study Chair — Childrens Hospital for Wales; Hans Merks, MD, PhD, Study Chair — Dutch Childhood Oncology Group
Locations (27):
- St. Anna Children's Hospital, Vienna, Austria
- Hopital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Vall d'Hebron University Hospital, Barcelona, Spain
- Uppsala University Hospital, Uppsala, Sweden
- University Children's Hospital, Zurich, Switzerland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Derived] Orbach D, Van Noesel MM, Brennan B, Corradini N, Alaggio R, Ben Arush M, Schoot RA, Berlanga P, Zanetti I, Hjalgrim LL, Di Corti F, Ramirez G, Casanova M, Ferrari A. Epithelioid hemangioendothelioma in children: The European Pediatric Soft Tissue Sarcoma Study Group experience. Pediatr Blood Cancer. 2022 Oct;69(10):e29882. doi: 10.1002/pbc.29882. Epub 2022 Jul 16. PMID 35841307
- [Derived] Schoot RA, Chisholm JC, Casanova M, Minard-Colin V, Geoerger B, Cameron AL, Coppadoro B, Zanetti I, Orbach D, Kelsey A, Rogers T, Guizani C, Elze M, Ben-Arush M, McHugh K, van Rijn RR, Ferman S, Gallego S, Ferrari A, Jenney M, Bisogno G, Merks JHM. Metastatic Rhabdomyosarcoma: Results of the European Paediatric Soft Tissue Sarcoma Study Group MTS 2008 Study and Pooled Analysis With the Concurrent BERNIE Study. J Clin Oncol. 2022 Nov 10;40(32):3730-3740. doi: 10.1200/JCO.21.02981. Epub 2022 Jun 16. PMID 35709412